CLINICAL TRIAL: NCT01137799
Title: A Double-Blind, Placebo-Controlled, Randomized, Four-Way Cross-Over Study To Investigate Effect Of Single Oral Doses Of JNJ-39393406 On Event-Related Potentials In Subjects With Stable Schizophrenia
Brief Title: The Effect of JNJ-39393406 on Event Related Potentials in Stable Schizophrenic Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Efficacy signals were insufficiently strong to justify recruitment of additional patients.
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016762
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Schizophrenia; Alzheimer's Disease; Cognition Disorders
Keywords: symptomatic treatment; cognition; cognitive deficits; schizophrenia; Alzheimer's Disease
MeSH Terms: conditions — Schizophrenia; Alzheimer Disease; Cognition Disorders | interventions — JNJ-39393406

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 001 (Experimental): JNJ-39393406 10mg nanosuspension (sort of liquid formulation) once daily (single dose)
  Interventions: Drug: JNJ-39393406
- 002 (Experimental): JNJ-39393406 30mg nanosuspension (sort of liquid formulation) once daily (single dose)
  Interventions: Drug: JNJ-39393406
- 003 (Experimental): JNJ-39393406 50mg nanosuspension (sort of liquid formulation) once daily (single dose)
  Interventions: Drug: JNJ-39393406
- 004 (Experimental): JNJ-39393406 100mg nanosuspension (sort of liquid formulation) once daily (single dose)
  Interventions: Drug: JNJ-39393406
- 005 (Experimental): JNJ-39393406 200mg nanosuspension (sort of liquid formulation) once daily (single dose)
  Interventions: Drug: JNJ-39393406
- 006 (Placebo Comparator): placebo Once daily (single dose)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: JNJ-39393406 — 50mg nanosuspension (sort of liquid formulation) once daily (single dose)
  Arms: 003
Drug: placebo — Once daily (single dose)
  Arms: 006
Drug: JNJ-39393406 — 200mg nanosuspension (sort of liquid formulation) once daily (single dose)
  Arms: 005
Drug: JNJ-39393406 — 100mg nanosuspension (sort of liquid formulation) once daily (single dose)
  Arms: 004
Drug: JNJ-39393406 — 10mg nanosuspension (sort of liquid formulation) once daily (single dose)
  Arms: 001
Drug: JNJ-39393406 — 30mg nanosuspension (sort of liquid formulation) once daily (single dose)
  Arms: 002

SUMMARY:
This study in patients with stable schizophrenia will investigate the effect of JNJ-39393406 on Event Related Potentials (Auditory Evoked Potential [AEP] P50, AEP P300 and Mismatch Negativity [MMN]) after single dose administration.

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor patient knows the name of the assigned drug), placebo-controlled, randomized (study drug assigned by chance), four-way-crossover trial (participants may receive different interventions sequentially during the trial) in patients with stable schizophrenia. The four-way-crossover treatment phase will consist of four blinded treatment periods separated by a wash out period (the period allowed for the entire administered drug to be eliminated from the body) of 6 to 14 days. The study duration for each patient will be approximately 12 weeks. Each patient enrolled will receive 3 (out of 5) dose levels of JNJ-39393406 and one dose of placebo. Part A of the study will include smoking patients with schizophrenia and will precede part B which will include non-smoking patients with schizophrenia. Safety evaluations include adverse event monitoring, vital signs and clinical laboratory tests. The study drug will be given as a single dose on Day 1 of each treatment period as a kind of liquid formulation with 240 mL non-carbonated water between 7:00 AM and 10:30 AM. Before dosing patients will be given a standard breakfast. The proposed dose levels for this study (Part A and Part B) will range from 10 to 200 mg.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 55 years of age, inclusive
* A known history of schizophrenia of at least 12 months by the referring psychiatrist
* DSM-IV criteria for Schizophrenia (including all subtypes)
* Stable treatment for at least 3 months (minor changes are acceptable upon confirmation by the sponsor representative)
* Medically stable on the basis of physical examination, medical history, vital signs, and 12-lead ECG performed at screening. If there are abnormalities, they must be consistent with the underlying illness in the study population
* Medically stable on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the subject may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the subject source documents and initialed by the investigator
* BMI between 18 and 35 kg/m² inclusive (BMI = weight/height²)
* For the pharmacogenomic component of this study subjects must have signed a separate written informed consent indicating willingness to participate in Part 1 genetic testing (mandatory), and indicate either consent or refusal for Part 2 DNA storage. Subject participation in the genetic testing component of the study (Part 1) is mandatory. Participation in the DNA storage component (Part 2) is voluntary and refusal to participate will not result in ineligibility for the main part of the study

Exclusion Criteria:

* A DSM-IV axis I diagnosis other than schizophrenia
* Clinically significant abnormal values for clinical chemistry, hematology or urinalysis at screening or admission. It is expected that laboratory values will generally be within the normal range for the laboratory, though minor deviations, which are not considered to be of clinical significance to the investigator, are acceptable. Values of ALT/AST < 2 fold the upper limit of normal will be allowed
* Clinically significant abnormal physical examination, vital signs or 12 lead ECG at screening. Minor deviations in ECG, which are not considered to be of clinical significance to the investigator, are acceptable
* QTcb >470ms
* A DSM-IV diagnosis of substance dependence within 6 months prior to screening evaluation (caffeine dependence is not exclusionary. Patients with a positive drug screen at screening may be included provided use does not lead to a DSM-IV diagnosis of substance dependence and patients consents to abstain from illegal drugs within 3 days prior to Day -1 and at any time during the study)
* Treatment-resistant subjects (failure to respond to two different antipsychotic drugs in the past)
* PANSS scores > 70
* Suicidal risk (assessed by the investigator such as, prior attempts to suicide, command hallucinations and / or hopelessness)
* Use of clozapine within 3 months before screening until follow-up
* Use of more than two antipsychotic drugs within 3 months before dosing until follow up

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2009-08; Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Improvement of deficits (i.e. sensory gating deficits) in event related potentials like Auditory Evoked Potentials P50 and P300 and Mismatch Negativity. | Predose and 2 and 5 hours post dose during each treatment period.

SECONDARY OUTCOMES:
Improvement in continuous performance testing | Predose, 2h and 5 post dosing during each treatment period
Plasma concentrations of JNJ-39393406 (PK blood samples) | Predose, 1h, 1h45, 3h, 4h45 and 6h postdose during each treatment period
Number of patients with clinical significant changes in vitals signs | Baseline, predose and 6h post dose during each treatment period and follow up visit.
Number of patients with clinical significant changes in ECG parameters | baseline, predose and 6h post dose during each treatment period and follow up
Number of patients with clinical clinical significant changes in clinical laboratory parameters | baseline, predose and 6h post dose during each treatment period and Follow Up

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.
Locations (4):
- Germany (4):
  - Berlin
  - Erlangen
  - München
  - Neuss

REFERENCES:
- [Derived] Winterer G, Gallinat J, Brinkmeyer J, Musso F, Kornhuber J, Thuerauf N, Rujescu D, Favis R, Sun Y, Franc MA, Ouwerkerk-Mahadevan S, Janssens L, Timmers M, Streffer JR. Allosteric alpha-7 nicotinic receptor modulation and P50 sensory gating in schizophrenia: a proof-of-mechanism study. Neuropharmacology. 2013 Jan;64:197-204. doi: 10.1016/j.neuropharm.2012.06.040. Epub 2012 Jul 2. PMID 22766391